CLINICAL TRIAL: NCT04863053
Title: Comparison of Serum Thromboxane B2 and Platelet Function Testing With the Multiplate® Device as Measures of Aspirin Resistance in Hong Kong Chinese Patients With Increased Cardiovascular Risk With Stable Coronary Heart Disease
Brief Title: Thromboxane B2 and Platelet Function Testing as Measures of Aspirin Resistance in Hong Kong Chinese Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Tomlinson, Professor, Chinese University of Hong Kong
Other Study IDs: ASPR
Record Dates: First submitted 2021-04-16; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood samples will be obtained from patients immediately before and 1 hour after aspirin dose after at least 10 h fast in the study centre. Blood samples obtained in lithium heparin tube for platelet aggregation test with Multiplate® analyzer will be sent for analysis immediately after blood collection. A 10 ml blood sample obtained in EDTA tube will be used for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable CHD patient: Patients aged ≥ 18 years who have a history of stable coronary heart disease (CHD) receiving long-term mono-antiplatelet therapy with aspirin (80 mg once daily)
  Interventions: Other: Blood samples will be taken to assess platelet function. There is no change in treatment.

INTERVENTIONS:
Other: Blood samples will be taken to assess platelet function. There is no change in treatment.

SUMMARY:
The hypotheses of the study are that the diagnostic accuracy of Multiplate® device for diagnosis of aspirin resistance is comparable to the serum TXB2 assay and that certain genetic polymorphisms and phenotypic factors significantly influence the antiplatelet effect of aspirin and contribute to aspirin resistance observed in this study.

DETAILED DESCRIPTION:
Fasting blood samples will be obtained from patients in the study centre after fasting overnight for at least 10 hours immediately before and 1 hour after the 80 mg aspirin dose. A 5-ml blood sample will be obtained in a serum separator tube and allowed to clot at room temperature followed by centrifugation at 4 degrees C. Separated serum will be stored in aliquots at -80°C until analysis of TXB2. A 3-ml blood sample will be obtained in a hirudin blood tube for the platelet aggregation test with the Multiplate® analyzer which will be performed within 3 hours after blood collection. A 10 ml blood sample will be obtained in an ethylene diamine tetra acetic acid (EDTA) tube to be used for DNA extraction. During the study, a total of 26 ml blood will be taken from each participant. Morning urine samples before and 1 hour after aspirin ingestion will also be collected and stored at -80 °C until measurement.

The platelet activity of the samples will be measured with the hirudin blood using the Multiplate analyzer from Roche (Roche Diagnostics International Ltd, CH-6343 Rotkreuz, Switzerland) according to the manufacturer's instructions for the arachidonic acid induced platelet aggregation (ASPI) test. It will be analyzed within 0.5-3 hours after blood collection.

The serum samples will be assayed for TXB2 with EIA kits from Cayman (Item no. 501020, Cayman Chemical, MI, USA) according to the manufacturer's instructions.

The urine will be assayed for 11-dehydro TXB2 using the enzyme-linked immunosorbent assay (EIA) kit from Cayman (Item no. 519510, Cayman Chemical, MI, USA) according to the manufacturer's instructions. The data will then be standardized with urinary creatinine measured with Cayman creatinine (urinary) colorimetric assay kit (item no 500701).

The 11-dehydro TXB2 data will be standardized with the urinary creatinine levels measured by Creatinine (urinary) Colorimetric Assay kit from Cayman (Item no. 500701, Cayman Chemical, MI, USA) according to the manufacturer's instructions.

Genomic DNA of the patients will be extracted from EDTA blood by using phenol chloroform. The following six single nucleotide polymorphisms (SNPs) will be investigated initially: ITGA2 rs1126643, ITGA2B rs5911, PTGS1 rs1330344, ADK rs16931294, PEAR1 rs12041331 and COX2 rs20417. The SNPs will be assayed with TaqMan SNP genotyping assays from Applied Biosystems (Applied Biosystems, Foster City, CA, USA) by Thermo Fisher Scientific according to the product inserts.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years who have a history of stable CHD receiving long-term mono-antiplatelet therapy with aspirin (80 mg once daily) for reducing cardiovascular risk will be recruited from the outpatient clinic.

Exclusion Criteria:

* Patients who are currently taking ticlopidine, clopidogrel, dipyridamole or other antiplatelet / antithrombotic agents will not be recruited.
* Patients who are on regular therapy with anti-inflammatory drugs, or others drugs containing aspirin or non-steroid anti-inflammatory drugs (NSAIDS), or traditional Chinese medicine that have direct effects on the haemostatic system, such as angelica, danshen, garlic, ginger, ginkgo and motherwort will not be included unless they are willing to stop these treatments for at least 2 weeks
* Patients will not be recruited if they had MI, stroke, coronary artery bypass surgery or other revascularization procedure, unstable angina or angioplasty within 3 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years who have a history of stable CHD receiving long-term mono-antiplatelet therapy with aspirin (80 mg once daily)
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
serum thromboxane B2 (TXB2) concentrations | Through study completion, an average of 1 year.
  Serum TXB2 concentrations will be measured by using an enzyme immunoassay kit to assess the adequacy of platelet cyclooxygenase (COX)-1 inactivation by aspirin. Each subject will only attend on one day.

SECONDARY OUTCOMES:
Multiplate® analyzer aspirin assay (ASPI test) platelet aggregation test | Through study completion, an average of 1 year.
  Multiplate® analyzer aspirin assay (ASPI test) platelet aggregation test will be measured by impedance aggregometry using the Multiplate® analyzer. Whole blood aggregation is performed using the on screen Multiplate protocol. Each subject will only attend on one day.
Genotyping of COX1 gene, which may be related to aspirin antiplatelet effect. | Through study completion, an average of 1 year.
  The COX1 gene polymorphism will be determined to assess if it is related to the aspirin antiplatelet effect measured by the ASPI test.
Genotyping of thromboxane A2 receptor (TBXA2R) gene, which may be related to aspirin antiplatelet effect. | Through study completion, an average of 1 year.
  The TBXA2R gene polymorphisms will be determined to assess if it is related to the aspirin antiplatelet effect measured by the ASPI test.

CONTACTS AND LOCATIONS:
Overall Officials: BRIAN TOMLINSON, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong